CLINICAL TRIAL: NCT04774510
Title: Optimized C-arm Cone Beam CT (CBCT) in the Neuro Angio-suite (NAS) for the Endovascular Treatment (EVT) of Acute Ischemic and Hemorrhagic Stroke
Brief Title: Optimized C-arm Cone Beam CT for the Endovascular Treatment (EVT) of Acute Stroke
Acronym: ASO-AVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210221
Record Dates: First submitted 2021-02-15; First posted 2021-03-01 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Stroke, Acute
Keywords: Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optimized C-ARM CBCT (Other): An optimized C-arm CBCT evaluation with a different acquisition geometry and a novel software for the rapid, quality improved and less-artefacts assessment of brain parenchyma and angiogram.
  Interventions: Other: Diagnostic Test: optimized C-Arm Cone Beam Computed Tomography

INTERVENTIONS:
Other: Diagnostic Test: optimized C-Arm Cone Beam Computed Tomography — Optimized C-ARM CBCT using new geometry and a novel software can rapidly and accurately detected brain abnormalities and hemorrhagic complications for critical patients with acute stroke. This rapid assessment would eliminate the need for the patient to be imaged in another scanner and be subsequently transported again to another room; all anatomic and physiologic imaging would occur in the neuro angiography suite (NAS).
  Other Names: C-ARM CBCT, XperCT Butterfly

SUMMARY:
When it comes to acute stroke, everyone deserves the best care. Today, more patients can benefit from endovascular treatment (EVT) in a comprehensive stroke center. With the significant advances in C-arm Cone Beam CT (CBCT) imagings directly in the neuro angio-suite (NAS), the investigators are now able to identify, plan and treat stroke patients in the NAS, without the need for a separate CT scan. This provides valuable, time-saving support for critical patients in acute need of EVT. The main objective is to assess the diagnostic confidence of this optimized C-arm Cone Beam CT, named in french ASO, in the NAS for the detection of brain abnormalities and hemorrhagic complications for critical patients with acute stroke. The secondary objectives are to study the variability of the diagnostic accuracy concerning the staging of the stroke, the analysis of the brain vessel, the relevance of artefact reduction post treatment and the amount of dose for this ASO.

DETAILED DESCRIPTION:
Design: ASO-AVC is a french academic pilot study by exploring the diagnostic confidence of optimized C-arm Cone Beam CT (ASO) realized directly in the neuro angio-suite (NAS).

To compare the effectiveness and safety of ASO diagnostic, the variability of the diagnostic accuracy concerning the staging of the stroke, the analysis of the brain vessel, the relevance of artefact reduction post treatment and the amount of delivered dose, the investigator proposed to assess clinical usefulness of ASO in the diagnostic process of stroke.

Intervention: No modification of patient care will be required by this protocol.

All patients participating in the study will undergo standard diagnostic, procedural and control imagings, which consist of : diagnostic imaging studies (MRI or CT scan), usual C-arm Cone Beam CT in the NAS during EVT to insure no procedural complication and control imaging studies (MRI or CT scan) at 24 hours ; decisions concerning further diagnostics will be made by the physician in charge.

Apart from theses standard imagings, patients will undergo the ASO. The ASO imagings will be anonymized and recorded in a centralized database called PACS (Picture Archiving and Communication System), in order to a centralized radiological reading by the Imaging Core Lab. They will be reviewed by radiologist readers to rate diagnostic image quality through a questionnaire, and in a second time the data will be included in a comparative evaluation with the diagnostic and control imagings.

ELIGIBILITY:
Inclusion Criteria:

aged ≥ 18 years diagnosed with an acute stroke and needed for a EVT affiliation to compulsory French social security scheme (beneficiary or right-holder) Consent from the patient if their level of consciousness is sufficient or from their relatives. If none is possible at the inclusion, consent will be obtained as soon as possible

Exclusion Criteria:

Being under tutelage or legal guardianship ; Ongoing pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
diagnostic confidence | baseline
  To assess the diagnostic confidence of ASO diagnostic with a centralized radiological reading

SECONDARY OUTCOMES:
Assess the degree of inter-observer agreement | baseline
  measuring assessor agreement in term of image quality and interpretation of ASO
Evaluate diagnostic agreement with conventional diagnostic imaging: MRI and CT scan | through study completion, an average of 48 hours
  Comparative evaluation with the diagnostic and control imagings.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa CHALUMEAU, MD, Principal Investigator — APHP
Locations (1):
- service de Neuroradiologie interventionnelle NEURI - Hôpital Bicêtre, Le Kremlin-Bicêtre, Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No